CLINICAL TRIAL: NCT02130232
Title: Appropriate Gestational Weight Gain in Overweight/Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CN-13-1628; 5R01HD073572-02 (NIH)
Record Dates: First submitted 2014-04-30; First posted 2014-05-05 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Gestational Weight Gain
Keywords: Gestational weight gain; Lifestyle; Intervention
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Intervention (Experimental): The goal of the intervention is to help women achieve the lower bound of the GWG range recommended by the Institutes of Medicine (IOM) for a given prepregnancy BMI category (i.e., 11 lbs for obese women and 15 lbs for overweight women). The pregnancy lifestyle intervention will be delivered by trained study dieticians via individual counseling sessions: 2 in-person and 11 telephone sessions delivered on a weekly basis, followed by telephone sessions delivered every other week through the end of pregnancy.
  Interventions: Behavioral: Lifestyle Intervention
- Usual Care (Active Comparator): Usual Medical Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Lifestyle Intervention
  Arms: Lifestyle Intervention
Other: Usual Care
  Arms: Usual Care

SUMMARY:
The goal of this trial is to investigate the efficacy of a lifestyle intervention of healthy diet and physical activity for helping overweight/obese pregnant women to achieve appropriate gestational weight gain (GWG) for their prepregnancy body mass index (BMI). The goal of the intervention is to help women achieve the lower bound of the GWG range recommended by the Institutes of Medicine (IOM) for a given prepregnancy BMI category (i.e., 11 lbs for obese women and 15 lbs for overweight women). The lifestyle intervention will be delivered via 2 in-person counseling sessions and 11 telephone contacts with study dieticians trained in motivational interviewing techniques. The lifestyle intervention will be compared to usual medical care. Outcomes will be assessed by trained study personnel at approximately 10 weeks and 32 weeks gestation, within several days of delivery and at 6 months and 12 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Pregravid BMI 25 to <40 (as determined from a measured pregravid weight in electronic medical record)

Exclusion Criteria:

* Diabetes
* Cardiovascular disease
* Gastrointestinal disease
* Bariatric surgery
* Lung disease
* Thyroid disease
* Eating disorder
* Cancer
* Bed rest or Gestational Diabetes in the current pregnancy
* Planning to get pregnant again or move within 1 year of delivery
* Substance abuse
* Serious mental health disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 398 (Actual)
Dates: Start 2014-04; Primary Completion 2019-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Rate of gestational weight gain per week | From pre-pregnancy weight to last pregnancy weight up to 21 weeks to 42 weeks of pregnancy
Proportion of women exceeding the Institute of Medicine's recommendation for rate of gestational weight gain per week | from pre-pregnancy weight up to 21 weeks to 42 weeks of pregnancy

SECONDARY OUTCOMES:
Total gestational weight gain | from pre-pregnancy weight to last pregnancy weight up to 24 weeks to 42 weeks
Proportion of women exceeding the Institute of Medicine's recommendation for total gestational weight gain per week | From pre-pregnancy weight to last pregnancy weight up to 24 weeks to 42 weeks
Rate of gestational weight gain between study clinical assessments | Rate of gestational weight gain between approximately 10 weeks and 32 weeks gestation (kilograms per week)
Diet - total calories from fat | Change in total calories from fat between study clinical assessments in pregnancy between 10 weeks and 32 weeks gestation
Diet - proportion of calories from fat | Change in proportion of calories from fat between study clinical assessments in pregnancy between 10 weeks and 32 weeks gestation
Physical Activity | Change in physical activity between study clinical assessments in pregnancy (i.e., between 10 weeks and 32 weeks gestation, approximately)
Metabolic marker - glycemia | Change in glucose between study clinical assessments in pregnancy (i.e., between 10 weeks and 32 weeks gestation, approximately)
Metabolic marker - insulinemia | Change in insulin between study clinical assessments in pregnancy (i.e., between 10 weeks and 32 weeks gestation, approximately)
Metabolic marker - lipids | Change in lipids between study clinical assessments in pregnancy (i.e., between 10 weeks and 32 weeks gestation, approximately)
Metabolic marker - leptin | Change in leptin between study clinical assessments in pregnancy (i.e., between 10 weeks and 32 weeks gestation, approximately)
Metabolic marker - adiponectin | Change in adiponectin between study clinical assessments in pregnancy (i.e., between 10 weeks and 32 weeks gestation, approximately)

CONTACTS AND LOCATIONS:
Overall Officials: Assiamira Ferrara, MD PhD, Principal Investigator — Kaiser Permanente Division of Research
Locations (2):
- United States (2):
  - Kaiser Permanente Oakland Medical Center, Oakland, California
  - Kaiser Permanente Santa Clara Medical Center, Santa Clara, California

REFERENCES:
- [Derived] Jake-Schoffman DE, Brown SD, Baiocchi M, Bibeau JL, Daubenmier J, Ferrara A, Galarce MN, Hartogensis W, Hecht FM, Hedderson MM, Moran PJ, Pagoto SL, Tsai AL, Waring ME, Kiernan M. Methods-Motivational Interviewing Approach for Enhanced Retention and Attendance. Am J Prev Med. 2021 Oct;61(4):606-617. doi: 10.1016/j.amepre.2021.04.005. PMID 34544560
- [Derived] Ferrara A, Hedderson MM, Brown SD, Ehrlich SF, Tsai AL, Feng J, Galarce M, Marcovina S, Catalano P, Quesenberry CP. A telehealth lifestyle intervention to reduce excess gestational weight gain in pregnant women with overweight or obesity (GLOW): a randomised, parallel-group, controlled trial. Lancet Diabetes Endocrinol. 2020 Jun;8(6):490-500. doi: 10.1016/S2213-8587(20)30107-8. PMID 32445736
- [Derived] Brown SD, Hedderson MM, Ehrlich SF, Galarce MN, Tsai AL, Quesenberry CP, Ferrara A. Gestational weight gain and optimal wellness (GLOW): rationale and methods for a randomized controlled trial of a lifestyle intervention among pregnant women with overweight or obesity. BMC Pregnancy Childbirth. 2019 Apr 30;19(1):145. doi: 10.1186/s12884-019-2293-8. PMID 31039753